CLINICAL TRIAL: NCT00001060
Title: A Phase I Trial of HIV-1 C4-V3 Polyvalent Peptide Vaccine in HIV-1 Infected Persons
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Lederle-Praxis Biologicals (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: DATRI 101; 11741 (Registry Identifier: DAIDS ES Registry Number); DATRI 0101
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; AIDS Vaccines; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

INTERVENTIONS:
Biological: HIV-1 C4-V3 Polyvalent Peptide Vaccine

SUMMARY:
To determine the safety of immunization with HIV-1 C4-V3 polyvalent peptide vaccine in HIV-infected persons. To determine the proportion of study participants immunized who develop new specificities or increased levels of neutralizing and other antibody responses, T-cell proliferative responses, and Class I restricted cytotoxic T-lymphocyte ( CTL ) responses.

HIV-1 C4-V3 polyvalent peptide vaccine contains amino acid sequences for selected epitopes from four of the most common HIV isolates in the United States and Europe, predicted to represent about 50-90 percent of the HIV isolates in the United States. It includes epitopes that generate potentially salutary immune responses and deletes epitopes that generate immune responses which might contribute to further immunopathogenesis.

DETAILED DESCRIPTION:
HIV-1 C4-V3 polyvalent peptide vaccine contains amino acid sequences for selected epitopes from four of the most common HIV isolates in the United States and Europe, predicted to represent about 50-90 percent of the HIV isolates in the United States. It includes epitopes that generate potentially salutary immune responses and deletes epitopes that generate immune responses which might contribute to further immunopathogenesis.

Patients are randomized to receive low-dose or high-dose HIV-1 C4-V3 polyvalent peptide vaccine in incomplete Freund's adjuvant (IFA), or IFA alone as control. Injections are administered on day 0 and at weeks 4, 8, 12, and 24. When patients entered at the lower vaccine dose (Cohort A) reach week 6, the data is reviewed and the higher dose cohort (Cohort B) will begin. When both cohorts reach week 14, data is evaluated and Cohort C begins vaccine administrations at a chosen vaccine dose. Within each cohort, eight patients receive vaccine plus IFA and two patients receive IFA alone. Patients are followed to week 52; 18 clinic visits and four telephone calls are required.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Other medically indicated vaccinations, provided they are administered at least 2 weeks before or after any study injection.
* Alcohol use limited to 1 oz per day of 100 proof.

Patients must have:

* HIV infection without evidence of AIDS.
* CD4 count > 500 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current evidence of underlying lung or liver disease.
* Suspected or diagnosed allergy to any vaccine component.
* Medical contraindication to protocol participation.
* Undergoing allergy skin testing or desensitization.

Concurrent Medication:

Excluded:

* Antiretroviral therapy (unless clinically indicated and with approval of investigator).
* Immunosuppressive or immunomodulatory therapy.
* Nonsteroidal anti-inflammatory agents (except short-term therapy for acute conditions).
* Drugs with known hepatotoxicity.
* Alcohol intake > 1 oz per day of 100 proof.

Patients with the following prior conditions are excluded:

* History of underlying lung disease.
* Abnormal chest radiograph within 2 weeks prior to first vaccine injection.
* History of underlying liver disease.
* Abnormal hepatitis B surface antigen or hepatitis C antibody test within 2 weeks prior to first vaccine injection.
* Abnormal liver function tests within 30 days prior to study entry.
* Evidence of uveitis by slit lamp exam within 2 weeks prior to study entry.
* Anergic as evidenced by negative skin test responses to all three antigens in a panel consisting of tetanus toxoid, mumps, and Candida albicans, within 6 weeks prior to first vaccine injection.
* Prior participation on an HIV vaccine trial.

Prior Medication:

Excluded within the past 3 months:

* Antiretroviral therapy.
* Immunosuppressive drugs.
* Alpha interferon or any immunomodulatory drugs.
* Any investigational HIV drugs or therapies. Current alcohol abuse.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bartlett JA, Study Chair; Tacket CO, Study Chair; Virani-Ketter N, Study Chair
Locations (1):
- Duke Univ Med Ctr, Durham, North Carolina, United States

REFERENCES:
- [Result] Bartlett JA, Wasserman SS, Hicks CB, Dodge RT, Weinhold KJ, Tacket CO, Ketter N, Wittek AE, Palker TJ, Haynes BF. Safety and immunogenicity of an HLA-based HIV envelope polyvalent synthetic peptide immunogen. DATRI 010 Study Group. Division of AIDS Treatment Research Initiative. AIDS. 1998 Jul 30;12(11):1291-300. doi: 10.1097/00002030-199811000-00010. PMID 9708408